CLINICAL TRIAL: NCT07329361
Title: Efficacy and Safety of Intra-articular Injections of Frozen Platelet-Rich Plasma in Patients With Knee Osteoarthritis: Randomized Control Trial
Brief Title: Efficacy and Safety of Intra-articular Injections of Frozen Platelet-Rich Plasma in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiKS Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCA-17/EC/25/CON
Record Dates: First submitted 2025-12-10; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frozen Platelet-Rich Plasma (Experimental)
  Interventions: Other: Platelet Rich Plasma
- Platelet-Rich Plasma (Active Comparator)
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Platelet Rich Plasma — Platelet-rich plasma stored by freezing
  Arms: Frozen Platelet-Rich Plasma
Other: Platelet Rich Plasma — Fresh Platelet-Rich Plasma
  Arms: Platelet-Rich Plasma

SUMMARY:
Evaluation of intra-articular injections in knee osteoarthritis using frozen-stored PRP. Compared with intra-articular injections of PRP applied at the time of collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Aged between 40 and 85 years old.
* Diagnosed with osteoarthritis through clinical radiological examination.
* Joint pain equal to or less than 75 points on the KOOS (pain).
* Radiological severity grades 1, 2, and 3 according to the Ahlbäck scale.
* Indication for intra-articular PRP infiltration.
* Body Mass Index values between 20 and 35.
* Negative serological tests for syphilis, HIV, HBV, and HCV.
* Possibility of observation during the follow-up period.
* Signature of informed consent.

Exclusion Criteria:

* Body mass index >35
* Diagnosed polyarticular disease.
* Previous arthroscopy in the last year.
* Severe mechanical deformity.
* Intra-articular hyaluronic acid injection in the last 12 months.
* Intra-articular corticosteroid or PRP injection in the last 6 months.
* Systemic autoimmune rheumatic disease (connective tissue diseases and systemic necrotizing vasculitis).
* Anemia or other hematological disorders.
* Positive serological tests for SYPHILIS, HIV, HBV, and HCV.
* Undergoing immunosuppressive treatments.
* Poorly controlled diabetes mellitus.
* Patients allergic to paracetamol.
* Pregnancy or breastfeeding.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
KOOS - Knee Injury and Osteoarthritis Outcome Score | 6 months
  From 0 (worst outcome) to 100 (best outcome)

SECONDARY OUTCOMES:
KOOS - Knee Injury and Osteoarthritis Outcome Score | 2 months
  From 0 (worst outcome) to 100 (best outcome)
VAS - Visual Analog Scale | 2 months
  From 0 (best outcome) to 10 (worst outcome)
VAS - Visual Analog Scale | 6 months
  From 0 (best outcome) to 10 (worst outcome)
Lequesne Index | 2 months
  A patient-completed questionnaire used to measure the severity of osteoarthritis assessing pain and function.
  From 0 (best outcome) to 24 (worst outcome)
Lequesne Index | 6 months
  A patient-completed questionnaire used to measure the severity of osteoarthritis assessing pain and function.
  From 0 (best outcome) to 24 (worst outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Arthroscopic Surgery Unit, MiKS Hosptial, Vitoria-Gasteiz, Araba/Álava, Spain